CLINICAL TRIAL: NCT04987073
Title: Preclinic Evaluation of a Vitamin D Analog in Vitamin D 24-hydroxylase Deficiency
Brief Title: Vitamin D Analog in Vitamin D 24-hydroxylase Deficiency
Acronym: VaraD-Cell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A03281-38
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Infantile Hypercalcemia - Severe Form
Keywords: CYP24A1; vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with CYP24A1 mutation (Experimental)
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — A skin biopsy to cultivate fibroblasts.

SUMMARY:
Preclinical evaluation of a vitamin D analog for the treatment of vitamin D 24-hydroxylase using fibroblast from patients with CYP24A1 mutation.

ELIGIBILITY:
Inclusion Criteria:

* biallelic mutation in CYP24A1
* consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Effects of the analog on vitamin D induced genes' expression | 3 years
  RNA quantification of genes induced by vitamin D in presence of analog in patients' fibroblast

CONTACTS AND LOCATIONS:
Locations (1):
- Arnaud Molin, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No